CLINICAL TRIAL: NCT03992911
Title: Phase II/III Trial of Simmtecan and 5-FU/LV Regimen (FOLFSIM) Plus Teripalimab Versus EP/EC in Advanced or Metastatic Neuroendocrine Carcinoma
Brief Title: Safety and Efficacy of FOLFSIM Plus Toripalimab in the Treatment of Advanced or Metastatic Neuroendocrine Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, MD, Professor, Chief of Department of GI Oncology, Peking University Cancer Hospital, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP-201
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Neuroendocrine Carcinoma of the Bladder
Keywords: Neuroendocrine Carcinoma; Simmtecan; Toripalimab
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Fluorouracil; toripalimab; PE regimen; EC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFSIM Plus Teripalimab (Experimental): Simmtecan and 5-FU/LV Regimen (FOLFSIM) Plus Teripalimab
  Interventions: Drug: Simmtecan, 5-FU and l-LV; Drug: Toripalimab
- EP/EC (Active Comparator): Etoposide plus Cisplatin or Carboplatin
  Interventions: Drug: Etoposide, Cisplatin; Drug: Etoposide, Carboplatin

INTERVENTIONS:
Drug: Simmtecan, 5-FU and l-LV — Simmtecan was administered intravenously at 80 mg per square meter on day1 with LV 400 mg per square meter administered as a 2-hour infusion, and 5-FU 2400 mg per square meter as a 46-hour infusion on day1 every 2 weeks in one course.
  Other Names: FOLFSIM regimen
  Arms: FOLFSIM Plus Teripalimab
Drug: Toripalimab — Toripalimab was administered intravenously at 240 mg on day 1 every 2 weeks in one course.
  Other Names: JS001
  Arms: FOLFSIM Plus Teripalimab
Drug: Etoposide, Cisplatin — Etoposide was administered intravenously at 100 mg per square meter on day 1,2,3 with Cisplatin at 80 mg per square meter on day 1 every 3 weeks in one course.
  Other Names: EP regimen
  Arms: EP/EC
Drug: Etoposide, Carboplatin — Etoposide was administered intravenously at 100 mg per square meter on day 1,2,3 and Carboplatin with AUC 5mg/mL/min on day 1 every 3 weeks in one course.
  Other Names: EC regimen
  Arms: EP/EC

SUMMARY:
This study is designed as Phase II/III. Phase II is aimed to evaluate safety and efficacy of Simmtecan and the 5-FU/LV regimen (FOLFSIM regimen) plus Toripalimab. Phase III is aimed to verify inferiority of the overall survival of FOLFSIM regimen plus Toripalimab in comparison with EP/EC in advanced or metastatic neuroendocrine cancer.

DETAILED DESCRIPTION:
This is a Phase II/III, randomized, two-part, multi-center study, in which subjects with advanced or metastatic neuroendocrine carcinoma will be enrolled.

This study will be conducted in two parts:

Part 1, the Phase II study was to: (i) evaluate the safety and tolerability of the FOLFSIM regimen plus Toripalimab; and (ii) identify the recommended dose; (iii) assess the antitumor activity; (iv) the pharmacokinetic (PK) parameters of the drugs in the regimen.

Part 2, the Phase III study was to verify inferiority of FOLFSIM regimen plus Toripalimab compared with the current standard chemotherapy (EP/EC regimen) in the first-line treatment of advanced or metastatic neuroendocrine carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed-consent form.
2. Male and Female aged between 18-75 years.
3. Histologically confirmed locally advanced or metastatic nonfunctional poorly-differentiated G3 neuroendocrine carcinoma(NEC), including small cell NEC, large cell NEC and MANEC.
4. Unresectable, including local advanced, recurrent or metastatic disease:

   Patients who had progressed after first-line platinum-based regimen or intolerance for treatment, or unwilling to receive current standard chemotherapy (only for phase II); Patients who has received no systemic chemotherapy, or relapsed at least 6 months since completion of adjuvant chemotherapy or radiotherapy.
5. At least 1 measurable lesion according to RECIST criteria;
6. Providing with tumor specimen (for testing the expression of PD L1 and the infiltrating lymphocytes);
7. Eastern Cooperative Oncology Group (ECOG) 0-1;
8. Adequate liver, kidney and bone marrow function; Screening laboratory values must meet the following criteria: hemoglobin ≥ 10.0 g/dL; neutrophils ≥ 1500 cells/ μL; platelets ≥ 100 x 10^3/ μL; total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1.5 x ULN, creatinine clearance >60ml/min (CockcroftGault equation), INR≤1.5, APTT≤1.5 x ULN;

Exclusion Criteria:

1. Histologically confirmed well differentiated G3 neuroendocrine tumor;
2. Evidence with active CNS disease or epilepsy;
3. Metastasis over 5 lesions;
4. Prior treatment with CPT-11 or antiPD1/PDL1/CTLA-4 antibody for neoadjuvant or adjuvant therapy;
5. Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix;
6. Predicted survival <3 months;
7. Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II NYHA, heart block >II grade, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm);
8. Any uncontrollable active infection, within past 1 week
9. Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism;
10. History with tuberculosis;
11. The side effects caused by the previous treatment of the subjects did not return to CTCAE ≤1; except hair loss and other tolerable events determined by investigator;
12. Hypersensitivity to Simmtecan or recombinant humanized antiPD1 monoclonal Ab or its components;
13. Prior antitumor therapy (including chemotherapy, target therapy, corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
14. Patients who received a potent inhibitor or inducer of CYP3A4 within 1 week prior to the first dose;
15. Prior radical radiothearpy within past 4 weeks;
16. Prior major surgery within past 4 weeks (diagnostic surgery excluded);
17. Prior live vaccine therapy within past 4 weeks;
18. Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml);
19. Pregnant or nursing;
20. Males or female of childbearing potential refuse to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 12 months after the last dose of study drug.
21. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Measure of time from study treatment to patient's death or lost to follow-up.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Measure of time from study treatment to disease progression or death.
Objective response rate | 2 years
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST)
Disease control rate | 2 years
  The sum of rates of partial response, complete response and steady disease based on Response Evaluation Criteria In Solid Tumors (RECIST).
Duration of response | 2 years
  Duration of Response by RECIST
The incidence of treatment related emergent adverse events（Safety and Tolerance) | 2 years
  Adverse reactions evaluation is based on the CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China